CLINICAL TRIAL: NCT05961761
Title: An Open Label Phase 2 Study on Propranolol and Pembrolizumab in Advanced Angiosarcoma and Undifferentiated Pleomorphic Sarcoma - a Scandinavian Sarcoma Group Collaboration
Brief Title: Propranolol and Pembrolizumab in Advanced Soft Tissue Sarcoma Patients
Acronym: PROPANE
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Niels Junker (Other)
Collaborators: Aarhus University Hospital (Other); Oslo University Hospital (Other); Karolinska University Hospital (Other)
Responsible Party: Sponsor-Investigator, Niels Junker, Consultant, MD, PhD, Principal Investigator, Herlev and Gentofte Hospital
Organization: Herlev and Gentofte Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SA2115
Record Dates: First submitted 2023-06-13; First posted 2023-07-27 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Soft Tissue Sarcoma Adult; Angiosarcoma; Undifferentiated Pleomorphic Sarcoma
Keywords: Immunotherapy; Propranolol; Pembrolizumab; PD-1 inhibitor; Sarcoma
MeSH Terms: conditions — Hemangiosarcoma; Histiocytoma, Malignant Fibrous; Sarcoma | interventions — Propranolol; pembrolizumab; spartalizumab

STUDY DESIGN:
Intervention Model Description: A Simon´s optimum two-stage design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Propranolol + pembrolizumab (Experimental): pembrolizumab 2 mg/kg every 3 weeks and propranolol 40 mg x2 daily until progression, unacceptable toxicity or patient withdrawal for a maximum of two years.
  Interventions: Drug: Propranolol; Drug: Pembrolizumab

INTERVENTIONS:
Drug: Propranolol — propranolol 40 mg x2 daily
  Other Names: Betablocker
Drug: Pembrolizumab — pembrolizumab 2 mg/kg every 3 weeks
  Other Names: anti PD-1

SUMMARY:
The goal of this phase 2 clinical trial is to test efficacy and tolerability of combining propranolol and pembrolizumab in patients with advanced angiosarcoma or undifferentiated pleomorphic sarcoma. The main questions aims to answer:

* Primary: determine the progression-free survival rate (PFSR) at 3 months

Secondary: determine the objective response rate (ORR), duration of Response (DOR), Progression Free Survival (PFS), Overall Survival (OS). Ensure the safety and tolerability, Determine Quality of Life (QoL)

• Exploratory: Characterize the TME

Participants will be asked to ensure

* Baseline biopsy and further optional biopsies
* Treatment propranolol 40 mg BID and pembrolizumab 2 mg/kg Q3 weeks
* Evaluation, blood counts, QoL and blood samples for biomarkers according to schedule

DETAILED DESCRIPTION:
Soft tissue sarcomas (STS) are mesenchymal derived tumors consisting of more than 50 subtypes, showing high metastatic features in approximately 50% of patients with intermediate and high-grade tumors. In spite of optimizing sequence of conventional systemic treatments with chemotherapy and tyrosine kinase inhibitors with an increase in overall survival from 12 to 18 months, the prognosis has not changed and is still a dismal 8% overall survival at 5 years. After four decades doxorubicin is still first line treatment as no new drugs has proven more effective and/or less toxic. Thus, new treatment modalities are needed.

Angiosarcomas (AS) and Undifferentiated Pleomorphic Sarcoma (UPS), comprising approximately 2% and 10% of STS respectively, are by definition high grade sarcomas characterized by an aggressive course. In the non-resectable advanced and metastatic setting treatment options are limited with short term palliative intent with median overall survival (OS) < 12 months. Patients are often elderly and with co-morbidities, increasing risk of severe toxicity from chemotherapy leading to significant deterioration of Quality of Life. New therapeutic options are needed.

Emerging results on immune modulating therapy with immune checkpoint inhibitors (ICI), have shown promising signals of potential benefit in certain subtypes of STS, especially in UPS and AS.

In tumors, neovascularization facilitate hypoxia, glucose deprivation and increased VEGF production leading to an immune suppressive tumor microenvironment (TME). This can in part be reverted by anti-angiogenic therapy including multitarget tyrosine kinase inhibitors. A proposed novel approach for targeting angiogenesis and potential immune modulatory mechanisms is through beta-adrenergic receptor (βAR) signaling. Preclinical data support combining βAR blockade with propranolol in combination with anti PD-1, and recently a phase 1 study showed the combination propranolol and pembrolizumab was well tolerated in melanoma patients.

This study is an open label, Simon two-stage single arm phase 2 study of pembrolizumab and propranolol in two separate cohorts. Patients will receive pembrolizumab 2 mg/kg every 3 weeks and propranolol 40 mg x2 daily until progression, unacceptable toxicity or patient withdrawal for a maximum of two years.

Up to 40 patients will be included in each separate cohort. Up to 18 patients in stage 1 and up to 22 patients in stage 2.

The primary objective is to determine progression-free survival rate (PFSR) at 3 months by Response Evaluation Criteria in Solid Tumors (RECIST v1.1)

The secondary objectives are to determine objective response rate (ORR) and duration of Response (DOR) using RECIST v 1.1, PFS and OS. Ensure safety and tolerability according to Common Terminology Criteria for Adverse Events (CTCAE version 5.0), and determine Quality of Life (QoL) using the 30 item European Organization for Research and Treatment of Cancer Quality of Life Questionnaire C30 (EORTC QLQ C30) questionnaire

The explorative objective is to characterize the TME, immune cells and markers both in tumors and in peripheral blood.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have signed and dated an IRB/IEC approved written informed consent form in accordance with regulatory and institutional guidelines. This must be obtained before the performance of any protocol related procedures that are not part of normal subject care
* Subjects must be willing and able to comply with scheduled visits, treatment schedule, laboratory testing, and other requirements of the study
* Histologically confirmed diagnosis of unresectable locally advanced or metastatic Angiosarcoma or Undifferentiated Pleomorphic Sarcoma, who has progressed/failed to provide clinical benefit on first line standard chemotherapy.
* Age ≥18 years
* Eastern Cooperative Oncology Group Performance Status (ECOG PS) score of ≤2 at the time of enrollment.
* Evaluable disease as defined by Response Evaluation Criteria in Solid Tumors (RECIST version 1.1).
* Available material from archived formalin-fixed paraffin-embedded tumor tissue obtained within 3 months of study enrollment for biomarker related studies. If not sufficient or available, a newly obtained core or excisional biopsy of a tumor lesion may be performed.
* Patients must have normal organ and marrow function as defined below:
* Absolute neutrophil count (ANC) ≥ 1 x 10⁹/L
* Platelet count ≥ 75 x 10⁹/L
* Serum bilirubin ≤ 1.5 x upper limit of normal (ULN) (patients with Gilbert's Syndrome must have a total bilirubin ≤ 50 mmol/L)
* Aspartate transaminase (AST)/Alanine transaminase (ALT) ≤ 5 x ULN
* Serum creatinine ≤ 1.5 x ULN or creatinine clearance (CrCl) ≥ 40 mL/min (using the Cockcroft-Gault formula)
* Women of childbearing potential (WOCBP): Agreement to use contraceptive methods with a failure rate of < 1 % per year during the treatment period and for at least 120 days after the treatment. Safe contraceptive methods for women are birth control pills, intrauterine device, contraceptive injection, contraceptive implant,contraceptive patch or contraceptive vaginal ring.
* Men who are sexually active with WOCBP must use any contraceptive method with a failure rate of less than 1% per year during the treatment period and for at least 120 days after the treatment.
* Women who are not of childbearing potential (ie, who are postmenopausal or surgically sterile) as well as azoospermic men do not require contraception

Exclusion Criteria:

* Have an anticipated life expectancy of <3 months.
* Moderate to severe degree of bronchial asthma or chronic obstructive pulmonary disease.
* Acute or non-stable congestive heart failure
* Any other condition listed as contraindication for treatment with propranolol according to SPC
* Have received any previous systemic therapy targeting the PD-1/PDL-1 signaling pathway or other immune checkpoint inhibitors.
* Have received propranolol within 4 weeks prior to treatment.
* Prior to study day one received radiation therapy, chemotherapy or targeted small molecule therapy within 2 weeks and/or monoclonal antibody treatment within 4 weeks.
* Not recovered from the effects of previously administered agents
* Clinically active or unstable CNS metastases as assessed by the treating physician
* Any serious or uncontrolled medical disorder that, in the opinion of the investigator, may increase the risk associated with study participation or study drug administration, impair the ability of the subject to receive protocol therapy, or interfere with the interpretation of study results
* Participants with active, known or suspected autoimmune disease. Participants with vitiligo, type I diabetes mellitus, residual hypothyroidism Inclusion criteria
* Subjects must have signed and dated an IRB/IEC approved written informed consent form in accordance with regulatory and institutional guidelines. This must be obtained before the performance of any protocol related procedures that are not part of normal subject care
* Subjects must be willing and able to comply with scheduled visits, treatment schedule, laboratory testing, and other requirements of the study
* Histologically confirmed diagnosis of unresectable locally advanced or metastatic Angiosarcoma or Undifferentiated Pleomorphic Sarcoma, who has progressed/failed to provide clinical benefit on first line standard chemotherapy.
* Age ≥18 years
* Eastern Cooperative Oncology Group Performance Status (ECOG PS) score of ≤2 at the time of enrollment.
* Evaluable disease as defined by Response Evaluation Criteria in Solid Tumors (RECIST version 1.1).
* Available material from archived formalin-fixed paraffin-embedded tumor tissue obtained within 3 months of study enrollment for biomarker related studies. If not sufficient or available, a newly obtained core or excisional biopsy of a tumor lesion may be performed.
* Patients must have normal organ and marrow function as defined below:
* Absolute neutrophil count (ANC) ≥ 1 x 10⁹/L
* Platelet count ≥ 75 x 10⁹/L
* Serum bilirubin ≤ 1.5 x upper limit of normal (ULN) (patients with Gilbert's Syndrome must have a total bilirubin ≤ 50 mmol/L)
* Aspartate transaminase (AST)/Alanine transaminase (ALT) ≤ 5 x ULN
* Serum creatinine ≤ 1.5 x ULN or creatinine clearance (CrCl) ≥ 40 mL/min (using the Cockcroft-Gault formula)
* Women of childbearing potential (WOCBP): Agreement to use contraceptive methods with a failure rate of < 1 % per year during the treatment period and for at least 120 days after the treatment. Safe contraceptive methods for women are birth control pills, intrauterine device, contraceptive injection, contraceptive implant,contraceptive patch or contraceptive vaginal ring.
* Men who are sexually active with WOCBP must use any contraceptive method with a failure rate of less than 1% per year during the treatment period and for at least 120 days after the treatment.
* Women who are not of childbearing potential (ie, who are postmenopausal or surgically sterile) as well as azoospermic men do not require contraception

Exclusion criteria

* Have an anticipated life expectancy of <3 months.
* Moderate to severe degree of bronchial asthma or chronic obstructive pulmonary disease.
* Acute or non-stable congestive heart failure
* Any other condition listed as contraindication for treatment with propranolol according to SPC
* Have received any previous systemic therapy targeting the PD-1/PDL-1 signaling pathway or other immune checkpoint inhibitors.
* Have received propranolol within 4 weeks prior to treatment.
* Prior to study day one received radiation therapy, chemotherapy or targeted small molecule therapy within 2 weeks and/or monoclonal antibody treatment within 4 weeks.
* Not recovered from the effects of previously administered agents
* Clinically active or unstable CNS metastases as assessed by the treating physician
* Any serious or uncontrolled medical disorder that, in the opinion of the investigator, may increase the risk associated with study participation or study drug administration, impair the ability of the subject to receive protocol therapy, or interfere with the interpretation of study results
* Participants with active, known or suspected autoimmune disease. Participants with vitiligo, type I diabetes mellitus, residual hypothyroidism due to autoimmune condition only requiring hormone replacement, psoriasis not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger are permitted to enroll.
* Participants with a condition requiring systemic treatment with either corticosteroids (>10 mg daily prednisone equivalents) or other immunosuppressive medications. Inhaled or topical steroids and adrenal replacement doses > 10 mg daily prednisone equivalents are permitted in the absence of active autoimmune disease.
* Patients should be excluded if they have known history of testing positive for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS)
* Allergies and Adverse Drug Reaction
* History of allergy to study drug components
* History of severe hypersensitivity reaction to any monoclonal antibody
* WOCBP who are pregnant or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2021-08-17 (Actual); Primary Completion 2028-01 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival rate | 3 months
  Determine the progression-free survival rate (PFSR) at 3 months by Response Evaluation Criteria in Solid Tumors (RECIST v1.1)

SECONDARY OUTCOMES:
Objective response rate | Approximately 6 months
  Determine the objective response rate (ORR) using RECIST v 1.1
Duration of Response | Up to 2 years
  Duration of Response (DOR) measured as time from response to progression according to RECIST v 1.1 or death.
Progression Free Survival | Up to 2 years
  Progression Free Survival (PFS) according to RECIST v 1.1
Overall Survival | Up to 2 years
  Overall Survival (OS).
Safety of the treatment | Up to 2 years
  Toxicity will be assessed by Adverse Events using Common Terminology Criteria for Adverse Events (CTCAE) v 5.0. Adverse events (AEs) of interest include any grade 3 or 4 treatment-related AEs leading to discontinuation.
  Safety is measured through the proportion of treated patients whose worst AEs of interest occurred within safety follow up after the last treatment.
Quality of Life assessment | Up to 2 years
  Determine Quality of Life (QoL) EORTC QLQ-C30

CONTACTS AND LOCATIONS:
Overall Officials: Niels Junker, MD, PhD, Principal Investigator — Herlev and Gentofte Hospital
Locations (4):
- Denmark (2):
  - Aarhus University Hospital, Aarhus
  - Herlev Gentofte Hospital, Herlev
- Oslo University Hospital, Oslo, Norway
- Karolinska University Hospital, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No